CLINICAL TRIAL: NCT05419609
Title: Office-based Limited Dissection SMAS Manipulation Under Local Anesthesia Versus Facility-based SMAS Manipulation: a Single-surgeon, Random-assignment Non-inferiority Study
Brief Title: Comparison of an Office-based Limited Facelift and Hospital-based Full Facelift
Acronym: COAL2
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dufresne, Craig, MD, PC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1278-8245
Record Dates: First submitted 2022-06-03; First posted 2022-06-15 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Skin Aging; Facial Asymmetry; Aging Problems
Keywords: Rhytidoplasty; Facelift; Rhytidectomy; Superficial Musculoaponeurotic System
MeSH Terms: conditions — Facial Asymmetry

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Office-based limited facelift (Experimental): Patients will undergo a limited facelift in the office. Patients will receive local anesthesia and optionally may receive an antianxiety medication.
  Interventions: Procedure: Limited facelift; Other: FACE-Q | Aesthetics - Satisfaction With Lower Face and Jawline; Other: FACE-Q | Aesthetics - Recovery Early Symptoms; Other: FACE-Q | Aesthetics - Satisfaction with Outcome; Other: FACE-Q | Aesthetics - Adverse Effects: Cheeks, Lower Face, Neck
- Hospital-based full facelift (Active Comparator): Patients will undergo a full facelift in the hospital or ambulatory surgical center. Patients will receive either general anesthesia or intravenous sedation.
  Interventions: Procedure: Full facelift; Other: FACE-Q | Aesthetics - Satisfaction With Lower Face and Jawline; Other: FACE-Q | Aesthetics - Recovery Early Symptoms; Other: FACE-Q | Aesthetics - Satisfaction with Outcome; Other: FACE-Q | Aesthetics - Adverse Effects: Cheeks, Lower Face, Neck

INTERVENTIONS:
Procedure: Limited facelift — A limited procedure under local anesthesia that addresses signs of aging in the lower face and neck
  Other Names: Limited dissection SMAS manipulation
  Arms: Office-based limited facelift
Procedure: Full facelift — A full face and neck lift that addresses signs of aging in the face and neck
  Other Names: SMAS manipulation
  Arms: Hospital-based full facelift
Other: FACE-Q | Aesthetics - Satisfaction With Lower Face and Jawline — Completed by patients. The FACE-Q | Aesthetics - Satisfaction With Lower Face and Jawline is a 5-item questionnaire. Each item is rated 1-4, with 1 being "Very Dissatisfied" and 4 being "Very Satisfied". Lower scores suggest the person may be less pleased with the appearance of their lower face and jawline.
Other: FACE-Q | Aesthetics - Recovery Early Symptoms — Completed by patients. The FACE-Q | Aesthetics - Recovery Early Symptoms is a 17-item questionnaire. Each item is rated 1-4, with 1 being "Not at all" and 4 being "Extremely". Lower scores suggest the person may be experiencing fewer symptoms early in their recovery following an aesthetic facial procedure.
Other: FACE-Q | Aesthetics - Satisfaction with Outcome — Completed by patients. The FACE-Q | Aesthetics - Satisfaction with Outcome is a 6-item questionnaire. Each item is rated 1-4, with 1 being "Definitely disagree" and 4 being "Definitely agree". Lower scores suggest the person may be less pleased with their final appearance following surgery and the decision to have an aesthetic facial procedure.
Other: FACE-Q | Aesthetics - Adverse Effects: Cheeks, Lower Face, Neck — Completed by patients. The FACE-Q | Aesthetics - Adverse Effects: Cheeks, Lower Face, Neck is a 15-item questionnaire. Each item is rated 1-3, with 1 being "Not at all" and 3 being "A lot". Lower scores suggest the person may be experiencing fewer chronic symptoms following an aesthetic facial procedure.

SUMMARY:
To compare safety, patient satisfaction, and technical correction between a limited and full facelift, patients meeting strict clinical and safety criteria for both types of facelift will be randomly assigned to have one of these procedures. In the context of this study, a limited facelift is done in the office under local anesthesia, and a full facelift is done in the hospital or ambulatory surgical center with either general anesthesia or intravenous sedation.

DETAILED DESCRIPTION:
While there are previous reports of facelift in an office-based setting without general anesthesia or intravenous sedation, these reports included patient demographic information, medical history, and complication rates only and did not compare their office-based facelift with a full facelift done in the hospital or ambulatory surgical center. Previous reports also included oral sedation for all patients.

The current study will address these gaps in what is known about office-based limited facelifts done with local anesthesia. Finally, the study will also ascertain patient satisfaction at 3 points-at the pre-operative visit, early post-operative visit, and final visit-using selected modules from the validated FACE-Q | Aesthetics survey.

ELIGIBILITY:
Inclusion Criteria:

* Patient willing to randomly undergo either a limited facelift done in the office or a full facelift done in the hospital
* Patient willing and able to accept financial responsibilities of undergoing either type of facelift.
* Patient able to provide informed consent
* Between age 40-years-old and 85-years-old
* No history of bleeding disorder
* BMI <25
* Stable weight
* Does not have implanted cardiac device
* Minimal anxiety
* No history of smoking
* Stable, good health
* Normal blood pressure or well-controlled hypertension
* Surgeon believes patient could tolerate and safely undergo either a limited facelift done in the office or a full facelift done in the hospital

Exclusion Criteria:

* Patient refusal to randomly undergo either a limited facelift done in the office or a full facelift done in the hospital
* Patient not willing or not able to accept financial responsibilities of undergoing either type of facelift.
* Patient unable to provide informed consent
* Under age 40-years-old or over 85-years-old
* History of bleeding disorder
* BMI >25
* Unstable weight
* Has implanted cardiac device
* Significant anxiety
* History of smoking
* Significant active disease (e.g., dementia, cancer, chronic respiratory illness, heart disease, etc.)
* Uncontrolled hypertension
* Surgeon believes patient could not tolerate or safely undergo either a limited facelift done in the office or a full facelift done in the hospital

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06-30 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Difference between groups in number of patients requiring treatment by surgeon for post-operative adverse effects | 1 hour following surgery and 2 weeks following surgery
  Post-operative adverse effects may be acute, such as hematoma or infection, or they may become apparent later, such as nerve injury. Not all post-operative adverse effects will require treatment, such as mild pain, swelling, or bruising.
Difference in post-operative aesthetic correction rating between groups | an average of 1 year following surgery
  Post-operative aesthetic correction rating is completed based on comparison with pre-operative photographs. Ratings possible are 1 (no improvement) to 5 (excellent).

SECONDARY OUTCOMES:
Change in score of "FACE-Q | Aesthetics - Satisfaction With Lower Face and Jawline" from baseline to last post-operative visit | an average of 30 days before surgery and again an average of 1 year following surgery
  The "FACE-Q | Aesthetics - Satisfaction With Lower Face and Jawline" is a validated patient satisfaction survey for the lower face and jawline.

OTHER OUTCOMES:
Difference of "FACE-Q | Aesthetics - Satisfaction With Lower Face and Jawline" baseline and last post-operative visit scores between groups | an average of 30 days before surgery and again an average of 1 year following surgery
  The "FACE-Q | Aesthetics - Satisfaction With Lower Face and Jawline" is a validated patient satisfaction survey for the lower face and jawline.
Difference of "FACE-Q - Recovery Early Symptoms" scores between groups | 1 week following surgery
  The "FACE-Q - Recovery Early Symptoms" is a validated patient satisfaction survey for the early post-operative period following aesthetic facial procedures.
Difference of "FACE-Q | Aesthetics - Satisfaction with Outcome" scores between groups | an average of 1 year following surgery
  The "FACE-Q | Aesthetics - Satisfaction with Outcome" is a validated patient satisfaction survey for final outcomes following aesthetic facial procedures.
Difference of "FACE-Q | Aesthetics - Adverse Effects: Cheeks, Lower Face, Neck" scores between groups | an average of 1 year following surgery
  FACE-Q | Aesthetics - Adverse Effects: Cheeks, Lower Face, Neck" is a validated patient satisfaction survey for chronic adverse post-operative events following aesthetic facial procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Craig R Dufresne, MD, Principal Investigator — Office of Dr Craig R Dufresne, MD, PC
Locations (1):
- Office of Craig R Dufresne, MD, PC, Fairfax, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
De-identified individual participant data (IPD) will not be available to other researchers.